CLINICAL TRIAL: NCT03232710
Title: A Single-dose, Two-treatment, Two-sequence, Two-period, Two Way Crossover Bioequivalence Study of Bosiqing Aripiprazole Orally Disintegrating Tablets and ABILIFY Under Fasting/Fed Condition
Brief Title: Bioequivalence Study of Bosiqing and ABILIFY Under Fasting/Fed Condition
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chengdu Kanghong Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: KH716-E01-CRP-1.1
Record Dates: First submitted 2017-07-24; First posted 2017-07-28 (Actual); Last update posted 2017-07-28 (Actual); Status verified 2017-07

CONDITIONS: Bioequivalence
MeSH Terms: interventions — Aripiprazole

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- pilot study group (Experimental)
  Interventions: Drug: abilify
- group 1 (under fasting condition) (Experimental)
  Interventions: Drug: Bosiqing; Drug: abilify
- group 2 (under fasting condition) (Experimental)
  Interventions: Drug: Bosiqing; Drug: abilify
- group 3 (under fed condition) (Experimental)
  Interventions: Drug: Bosiqing; Drug: abilify
- group 4 (under fed condition) (Experimental)
  Interventions: Drug: Bosiqing; Drug: abilify

INTERVENTIONS:
Drug: Bosiqing — Aripiprazole Orally disintegrating tablets 10mg
  Arms: group 1 (under fasting condition); group 2 (under fasting condition); group 3 (under fed condition); group 4 (under fed condition)
Drug: abilify — Aripiprazol orodispersible tablets 10mg

SUMMARY:
To compare the rate and extent of absorption of Aripiprazole Orally disintegrating tablets 10 mg of Chengdu Kanghong Pharmaceutical Group Co.,Ltd, China and ABILIFY (Aripiprazole) 10 mg orodispersible tablets of Otsuka Pharmaceutical Europe Ltd. in healthy, adult, human subjects under fasting/fed condition as well as to monitor the safety and tolerability of subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects willing to adhere to the protocol requirements and to provide written informed consent.
2. Subjects aged between 45 and 65 years，healthy male and non-pregnant, non breast feeding female.
3. Subjects' weight within clinically acceptable normal range according to normal values for Body Mass Index (19.00 to 26.00 kg/m2) with minimum of 50 kg weight for male, and minimum of 45 kg weight for female.
4. No medical history of significant cardiovascular, pulmonary, hepatic, renal, gastrointestinal, endocrine, immunological, dermatological, neurological, urogenital or psychiatric disease or disorder.

Exclusion Criteria:

* 1)Subjects with family history of muscular dystonia or the subject has had the drug source dystonia.

  2）Subject with history of a asthma. 3）Subject with any (acute or chronic) history of mental illness or have family history of mental illness.

  4）Subject have alzheimer's or alzheimer's disease. 5）Subject was hospitalized within 60 days prior to the first dose of the study drug 6）Subject smoking more than five cigarettes within 1 month prior to the first dose study drug.

  7）History or presence of significant easy bruising or bleeding 8）History or presence of drug abuse. 9）History of allergic reactions. 10）History or presence of taking psychotropic drugs。 11）Subjects having positive urine screen for drugs of abuse including Methamphetamine, MDMA, ketamine, morphine, heroin.

  12）Any treatment which could bring about induction or inhibition of hepatic microsomal enzyme system within 3 weeks prior to Period 01 dosing.

  13）Consumption of hypericum perforatum containing products and grapefruit or grapefruit juice from 72 hours prior admission to 3 days after trail end.

  14）Subject involved other clinical trials of drugs within 3 months prior to period 01 dosing.

  15）Subject with abnormal laboratory tests and diagnosed by physicians as clinically significant 17）Abnormal vital signs test for any one or more:

Abnormal blood pressure:

* Systolic pressure is lower than 80mmHg and/or diastolic pressure down to 40mmHg in sitting position.
* Systolic pressure is higher than 140mmHg and/or diastolic pressure higher than 90mmHg in sitting position.

Abnormal cardiac rate:

* cardiac rate lower than 50
* cardiac rate higher than 50 18）Blood alcohol test values≥10mg/dL 19）Volunteer who have donated blood components within 2 weeks prior to the first dose or donated blood (more than 200 ml within 4 weeks; more than 400 ml within 60 days) prior to the first dose; Volunteer who plan to donate blood during the study or 4 weeks after study; Volunteer who lost blood (more than 50ml within 7days or more than 400ml within 30 days) for surgery.

  20）Subjects not willing to follow approved birth control methods for the duration of the study 21）ubjects having positive Serum β-hCG test. 22）Subjects plan to donate sperm during study period or 30 days after study 23）Hamilton depression Rating Scale ( 17 ) score above 7 points. 24）History of blood phobia. Subjects whom the investigator deems necessary to exclude.

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2017-06-26 (Actual); Primary Completion 2018-04-30 (Estimated); Study Completion 2018-06-30 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetic parameter: Cmax | day 54
  Bioequivalence based on Peak Plasma Concentration (Cmax) under fasting and fed condition
Pharmacokinetic parameter: AUC | day 54
  Bioequivalence based on Area under the plasma concentration versus time curves (AUC) under fasting and fed condition

SECONDARY OUTCOMES:
Adverse Events | up to day 54
  To observe the type, incidence and severity of adverse events in the study.

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital of Sichuan University, Chengdu, Sichuan, China